CLINICAL TRIAL: NCT04213833
Title: Effect of Palatable Lidocaine Gel Versus Dexmedetomidine on Gag Reflex During Propofol Based Sedation for Patients Undergoing Elective Upper Gastrointestinal Endoscopy. A Randomized Controlled Study
Brief Title: Effect of Palatable Lidocaine Gel on Gag Reflex for Patients Undergoing Upper Gastrointestinal Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Shereen Elsayed Abd Ellatif, lecturer of anesthesia and surgical intensive care, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5788-31-12-2019
Record Dates: First submitted 2019-12-23; First posted 2019-12-30 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Gastro-Intestinal Disorder
Keywords: palatable lidocaine; dexmedetomidine; gag reflex; gastrointestinal endoscopy
MeSH Terms: conditions — Digestive System Diseases; Gagging | interventions — Propofol; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: participant and endoscopist
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group I (control group) (Placebo Comparator): patients will receive propofol 50 mg
  Interventions: Drug: Propofol Injection [Diprivan]
- group II (Active Comparator): patients will receive propofol 50 mg + dexmedetomidine 0.5 mcg/ kg
  Interventions: Drug: Dexmedetomidine [Precedex]
- group III (Active Comparator): patients will receive propofol 50 mg +15 g palatable lidocaine gel
  Interventions: Drug: Palatable Lidocaine Topical Gel

INTERVENTIONS:
Drug: Propofol Injection [Diprivan] — patients will be sedated with 50 mg propofol(10 mg/ml) given slowly intravenously over 1 min
  Arms: group I (control group)
Drug: Dexmedetomidine [Precedex] — patients will received 0.5 mcg/ kg dexmedetomidine intravenously followed by syringe containing 50 mg propofol(10 mg/ml).
  Other Names: propofol
  Arms: group II
Drug: Palatable Lidocaine Topical Gel — 15 g of palatable lidocaine gel will be gradually applied 3-5 min before the endoscopy at three consecutive 30-s intervals to the base of the tongue, the palate and the peritonsillar areas and the patients will be informed to spread it within their mouth with their tongue and swallow it later to cover the oropharynx and esophagus. Patients will be asked to register the onset of numbness, then patient will receive syringe containing 50 mg propofol (10 mg/ml) intravenously as a sedation.
  Other Names: propofol
  Arms: group III

SUMMARY:
* The development of upper gastrointestinal endoscopy (UGIE) has greatly expanded the diagnostic and therapeutic capabilities of gastroenterologists. The patient's tolerance to procedure and endoscopist's satisfaction increase when sedation is used along with topical pharyngeal anesthesia.
* Numerous agents are available for moderate sedation in endoscopy such as propofol, midazolam, ketamine, fentanyl and dexmedetomidine, the choice of a particular sedative agent depends on its availability, cost and experience of the endoscopist and patient with that sedative agent. However, these i.v. anesthetics may be associated with complications especially in elderly patients or in those with other comorbidities, as apnea, hypoxia, hypotension, and paradoxical agitation, in which the patient becomes agitated rather than sleepy from the sedation, leading to increased morbidity and the duration of the patient's hospitalization.
* Local application of lidocaine to the oral cavity and the oropharynx, will attenuate or even abolish the gag reflex increasing the patient's comfort thus decreasing the dose of i.v. anesthetics with their potential complications.
* Up to our knowledge, there is no study done to evaluate the effect of palatable lidocaine gel versus I .v dexmedetomidine on the incidence of gag reflex and total propofol consumption during elective upper gastrointestinal endoscopy.

DETAILED DESCRIPTION:
Upper gastrointestinal tract endoscopy (UGIE) is a valuable procedure that is commonly used for the diagnosis of possible causes of upper gastrointestinal tract (GIT) symptoms such as bleeding, pain, dysphagia, recurrent vomiting and reflux. Moreover, it is a safe and easy procedure for taking biopsy samples for suspected esophageal, gastric and duodenal diseases, grading and even ligating varices [1, 2].

UGIE is widely performed under propofol sedation that considered a safe sedation technique and alleviates the sympathetic response to the procedure. However, gag reflex and retching still exist in approximately 29% of those patients despite being under propofol sedation [3]. Any further trial of deepening sedation in order to minimize gagging may compromise hemodynamics and cause respiratory depression. These complications add to the overall costs as it increases morbidity and duration of patients' hospitalization. On the other hand, continued gag reflex could affect the safety of the procedure, patient's tolerance and endoscopist's satisfaction [4].

Dexmedetomidine, a short-acting selective α2-agonist, has been used frequently as a sedoanalgesic in many diagnostic and therapeutic procedures [5]. It provides unique sedative activity not present in conventional sedatives so it is unlikely to cause restlessness or respiratory depression was seen with Gaba aminobutyric acid (GABA) receptor agonists such as propofol. Therefore it minimizes physical and emotional distress and enhances successful completion of the procedure without remarkable gag reflex [6]. However, many clinicians may have qualms regarding the safety profile of dexmedetomidine usage in such endoscopic procedures due to its well known hemodynamic side effects (especially bradycardia and hypotension) [7].

Topical pharyngeal anesthesia(TPA) has been used to avoid such complications resulting from deepening sedation through increase i.v anesthetic doses of propofol or adjuvants that may be used as dexmedetomidine. TPA is preferred in many centers, particularly for diagnostic endoscopy [8, 9].

Lidocaine is widely used for TPA. The spray, gel and inhaler forms of it are commercially available. However, application of lidocaine gel to the oral cavity and the oropharynx, especially the base of the tongue, palate, uvula, palatopharyngeal, palatoglossal folds and posterior pharyngeal wall will attenuate or even abolish the gag reflex while introducing the UGIE, thus increasing the patient's comfort and tolerance to the procedure and decreasing the dose of i.v. anesthetics with their potential complications [10, 11].

Palatable lidocaine gel is a local anesthetic that stabilizes the neuronal membrane through hindering the ionic fluxes that initiate and transmit impulses, thereby giving a local anesthetic action. It is a safe, well-tolerated and quite promising TPA particularly in elderly patients and in patients with comorbidities in office-based endoscopy [12].

We hypothesize that the usage of topical palatable lidocaine gel may have an impact on decreasing the incidence of gag reflex and total propofol consumption during upper gastrointestinal endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patient acceptance. Age 21-60 years old of either sex. BMI < 30 kg/m2 ASA I and ASA II. scheduled for elective upper GIT endoscopy

Exclusion Criteria:

* History of clinically significant cardiovascular, respiratory diseases (as obstructive sleep apnea, severe COPD or asthma) History of psychiatric disease History of allergy to any of the study drugs

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Gag reflex | through endoscopic procedure up to one hour
  will be assessed as ''present or not" when a vomiting like response will provoked upon introduction of the endoscope.

SECONDARY OUTCOMES:
heart rate | every 2 min for the first 10 min of the procedure, then every 5 min till the end of the procedure.
  Intraoperative hemodynamics
mean blood pressure | every 2 min for the first 10 min of the procedure, then every 5 min till the end of the procedure.
  Intraoperative hemodynamics
Patient's satisfaction regarding discomfort (gagging and pain) | 2 hours post the procedure
  will be assessed using numerical rating scale from 1 to 10 (1=satisfied and tolerated well the procedure to 10=unsatisfied)
Endoscopist's satisfaction regarding gagging and difficulty of performing the procedure | through endoscopic procedure up to one hour
  using numerical rating scale from 1 to 10 (1=no gagging/difficulty to 10=maximum gagging/ difficulty)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, zagazig university, Zagazig, Elsharqya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
planned after the completion of the study and publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: planned after the completion of the study and publication
Access Criteria: contact of principal investigator

REFERENCES:
- [Background] Ghallab M, Hussien RM, Samir GM, Ibrhaim DA. Palatal lidocaine gel as an adjuvant to propofol versus propofol only for sedation during upper gastrointestinal tract endoscopy: a comparative study. Ain-Shams J Anesthesiol 2014; 7:524-9.
- [Background] Samson S, George SK, Vinoth B, Khan MS, Akila B. Comparison of dexmedetomidine, midazolam, and propofol as an optimal sedative for upper gastrointestinal endoscopy: A randomized controlled trial. Journal of Digestive Endoscopy 2014;5(2) :51-7.
- [Background] Ramsay MA, Savege TM, Simpson BR, Goodwin R. Controlled sedation with alphaxalone-alphadolone. Br Med J. 1974 Jun 22;2(5920):656-9. doi: 10.1136/bmj.2.5920.656. PMID 4835444
- [Background] Bassi GS, Humphris GM, Longman LP. The etiology and management of gagging: a review of the literature. J Prosthet Dent. 2004 May;91(5):459-67. doi: 10.1016/S0022391304000939. PMID 15153854
- [Background] Abbas I, Hassanein A, Mokhtar M. Effect of low dose ketamine versus dexmedetomidine on gag reflex during propofol based sedation during upper gastrointestinal endoscopy. A randomized controlled study. Egyptian Journal of Anaesthesia 2017;33: 165-70.
- [Result] Heuss LT, Hanhart A, Dell-Kuster S, Zdrnja K, Ortmann M, Beglinger C, Bucher HC, Degen L. Propofol sedation alone or in combination with pharyngeal lidocaine anesthesia for routine upper GI endoscopy: a randomized, double-blind, placebo-controlled, non-inferiority trial. Gastrointest Endosc. 2011 Dec;74(6):1207-14. doi: 10.1016/j.gie.2011.07.072. Epub 2011 Oct 13. PMID 22000794